CLINICAL TRIAL: NCT06680284
Title: Greening the Operating Room: Auditing Anesthesia Generated Wastes and Exploring Strategies to Reduce, Reuse and Recycle
Brief Title: Toronto Western Hospital (TWH) Waste Audit
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 21-6124
Record Dates: First submitted 2024-08-21; First posted 2024-11-08 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-03

CONDITIONS: Audit of Medical Waste Disposal
Keywords: Medical Waste; Waste; Waste Disposal; Anesthesia; Anesthesia Waste; Anesthesia Waste Disposal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Staff anesthesiologists or anesthesia fellows: Participating study subjects will go through a staff education program to encourage proper waste disposal.
  Interventions: Other: Staff Education Program

INTERVENTIONS:
Other: Staff Education Program — A staff education and environmental awareness campaign and in-service to highlight strategies to reduce, reuse, and recycle waste, as well as proper waste disposal practice, will be implemented by way of instructional posters, e-learning modules, a grand rounds presentation, journal club discussion, and brainstorming sessions for waste reduction, reuse and recycle and a brief knowledge test at the end.

SUMMARY:
The goal of this observational study is to learn about the amount and types of anesthesia wastes generated for each surgical case at the Toronto Western Hospital (TWH). The main questions it aims to answer are:

* The amount of anesthesia waste generated per surgical case at TWH
* The amount of wastes that are inappropriately discarded
* The percentage of discarded waste that can be reused or recycled
* The percentage of recyclable waste that is actually recycled
* The percentage of discarded waste that is appropriately sent to landfill
* The financial cost of waste disposal
* The impact of a staff education program on waste reduction and proper waste disposal

The research team will conduct the audit by inspecting the contents of the waste bins and bags following completion of a surgery.

DETAILED DESCRIPTION:
Environmental pollution by healthcare waste is a complex and pervasive problem. Canadian hospitals produce a staggering 300 tons of medical waste daily and ~30% of wastes are generated by surgery and anesthesia services. A quarter of the solid waste associated with surgery is likely to be of anesthesia origin, with plastics (e.g. face masks, breathing circuits and IV sets) forming almost half of the total anesthetic waste volume, and mostly being discarded in landfills. Not only do they pose serious environmental harm to wildlife, these plastics also pose health risk to humans. Because plastics are resistant to many natural processes of degradation, microplastics can persist in the environment for hundreds of years with the potential to contaminate and bioaccumulate up the food chains through agricultural soils and the water supply. The need for operating room (OR) greening initiatives is indeed desperately urgent.

Solid waste generated by anesthesia is classified as either general waste or medical / biohazardous waste. General waste includes papers, plastic disposables and packaging materials and clean general wastes are recyclable. Medical waste encompasses sharps, pharmaceuticals, and materials that are contaminated by blood or infectious materials. They are not recyclable and require expensive treatment (e.g., autoclave and incineration) prior to final disposal. Thus, proper understanding of the type of waste (i.e. medical vs. general, recyclable vs. non-recyclable) and awareness of proper waste management procedures is important to avoid improper waste segregation and unneeded expensive biohazardous processing.

Among all the waste management options, waste reduction is most important. This is followed by reuse / reprocessing to prolong the product life cycle. Recycling should be considered when 'reduce' and 'reuse' have been maximized, and can decrease the volume of waste sent to landfills. However, recent strict contamination limits on the importation of recyclable plastics, especially in China, have caused a major slowdown in global recycling. Additionally, a lack of institutional culture of environmental sustainability, a lack of knowledge of proper waste segregation and recycling, and concerns about the extra workload associated with sorting for plastic recycling are some of the major institutional and human barriers that impede waste reduction and proper disposal efforts. Fortunately, a staff education and improvement program can overcome these barriers.

Despite these environmental threats, there are few published studies on anesthesia waste or guidelines for anesthesia waste management. This study first aims to quantify the magnitude of anesthesia wastes generated in the Toronto Western Hospital (TWH) operating room, then implement a staff education and waste awareness program, and finally measure the impact of such an education program on waste reduction, reuse and recycling.

The study includes 6 phases.

i. Phase 1 (4 months): The planning phase to conduct meetings with Operating Room leadership and Environmental Services to plan for a general and medical waste collection system in the operating room for this study.

ii. Phase 2 (2 months): 1-week prospective collection of solid wastes for each type of surgical service at TWH without notifying anesthesia staff; the collection will continue for 5 consecutive working weekdays in 1 week.

iii. Phase 3 (2 month): Analysis of waste collection data and report to anesthesia staff.

iv. Phase 4 (3 months): Staff education and environmental awareness campaign and in-service to highlight the reduce, reuse and recycle concepts and proper waste disposal practice.

v. Phase 5 (2 months): Repeat 1-week collection of wastes for each type of surgical procedure.

vi. Phase 6 (1 month): A second analysis and report of waste generation and disposal to the Department of Anesthesia.

Data will be collected for a minimum of 10 cases for each surgical type of varying duration. Descriptive statistics will be used to describe surgical case volume during the study period. Two-sample Student's t-test will be used to compare the daily weight of general, medical and recyclable solid wastes between the baseline study period and the second assessment period after staff education. A P value < 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

• Must be an anesthesia staff, resident or an anesthesia assistant at Toronto Western Hospital.

Exclusion Criteria:

• Inability to give informed consent to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Anesthesia staff, residents and assistants within the Toronto Western Hospital.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Measure the amount of all types of anesthesia waste generated per surgical case at Toronto Western Hospital. | Average 14 months after the beginning of the study.
  Measure the amount of anesthesia waste (general waste and medical waste) generated on average per surgical case. All general and medical anesthesia waste will further be categorized into into plastic and non plastic, reusable and non-reusable, and recyclable and non-recyclable; all quantified by weight in kilograms.

SECONDARY OUTCOMES:
Measure the incidence of inappropriate waste disposal | Average 14 months after the beginning of the study.
  The incidence of inappropriate waste disposal i.e., general wastes into the medical waste bin and vice versa, and weight in kilograms of recyclables remaining within the general and infectious waste
Measure the incidence of reusable general wastes that is discarded at Toronto Western Hospital. | Average 14 months after the beginning of the study.
  Measure of the amount of non-contaminated, reusable general wastes that is inappropriately discarded, measured by the average number of occurrence per surgical case and quantified in percentage.
Measure the incidence of recyclable general wastes that is discarded at Toronto Western Hospital. | Average 14 months after the beginning of the study.
  Measure of the amount of non-contaminated, recyclable general wastes that is inappropriately discarded, measured by the average number of occurrence per surgical case and quantified in percentage.
The amount of soft plastic packaging waste generated per case that is discarded | Average 14 months after the beginning of the study.
  The amount of soft plastic packaging waste generated on average per surgical case, that is discarded to landfill; quantified by weight in kilograms
To see the impact of anesthesia staff education program on the waste management and disposal behavior and practices among the anesthesia staff at Toronto Western Hospital.. | Average 14 months after the beginning of the study.
  The amount of change by weight of the appropriately disposed anesthesia waste by the anesthesia staff per surgical case in the second audit from the first audit will reflect the impact of staff education campaign on the staff behavior and practices; quantified in percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Chan, MD, FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No